CLINICAL TRIAL: NCT07394335
Title: Large Language Model (LLM) as a Tutor in Urodynamic Education: A Prospective Learning Curve Study Among Urology Residents
Brief Title: LLM in Urodynamic Education
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huseyin Kocakgol (Other)
Responsible Party: Sponsor-Investigator, Huseyin Kocakgol, MD, Urology, Erzurum City Hospital
Organization: Erzurum City Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: URO-LLM-UDS-2026
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Urodynamic Interpretation Skills
Keywords: Urodynamic Education, Learning Curve, Urology Residency, Large Language Models Training, LLM

STUDY DESIGN:
Intervention Model Description: Participants undergo a single-arm, prospective educational intervention with repeated assessments (pre-test, mid-test, and post-test) to evaluate changes in urodynamic interpretation performance over time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LLM-Based Urodynamic Education (Experimental): Participants receive a structured urodynamic education program supported by a large language model acting as an interactive tutor.
  Interventions: Other: LLM-Based Urodynamic Tutoring

INTERVENTIONS:
Other: LLM-Based Urodynamic Tutoring — Participants receive a structured urodynamic education program supported by a large language model acting as an interactive tutor.
  Other Names: LLM-Based Urodynamic Education

SUMMARY:
Urodynamic investigations, including cystometry, pressure-flow studies, and electromyography, are considered the gold standard for the objective diagnosis of lower urinary tract dysfunction according to current international guidelines. However, accurate interpretation requires simultaneous analysis of multiple pressure signals, identification of artifacts, and application of complex nomograms, making urodynamics one of the most challenging diagnostic skills to master during urology residency training. Traditional training largely depends on apprenticeship-based exposure, which is highly variable across training centers. The primary aim of this prospective educational study is to evaluate the effectiveness of a large language model (LLM), as an interactive tutor in improving urology residents' urodynamic interpretation skills and learning curve. By providing structured theoretical instruction, case-based guidance, and real-time feedback through a standardized case pool, this study investigates whether AI-assisted mentorship can accelerate skill acquisition, enhance diagnostic accuracy, and offer a standardized, accessible educational model for urodynamic training.

DETAILED DESCRIPTION:
Urodynamic testing, including cystometry, pressure-flow studies, and electromyography, represents the gold standard for the objective evaluation of lower urinary tract dysfunction. Despite its clinical importance, urodynamic interpretation requires advanced analytical skills, including simultaneous assessment of vesical, abdominal, and detrusor pressures, recognition of technical artifacts, and application of established nomograms. Consequently, mastery of urodynamic interpretation during urology residency training remains challenging and highly dependent on variable case exposure and faculty availability.

This prospective, single-center educational study is designed to assess the effectiveness of a large language model (LLM) configured as an interactive educational tutor in improving urology residents' urodynamic interpretation skills and learning curve. The study aims to determine whether structured, AI-assisted mentorship can provide a standardized and scalable alternative to traditional apprenticeship-based training.

Eligible participants include urology residents without prior formal urodynamic course certification. The educational intervention utilizes a curated library of 45 fully anonymized urodynamic tracings performed in accordance with International Continence Society standards. These cases represent a balanced spectrum of normal findings and common urodynamic diagnoses, including bladder outlet obstruction, detrusor overactivity, and reduced bladder compliance. All cases are validated by experienced urologists prior to inclusion.

The training protocol consists of sequential phases: a baseline assessment (pre-test), structured theoretical instruction delivered via an LLM-based tutoring interface, supervised case analysis with artifact recognition, interactive mentored interpretation, an intermediate assessment (mid-test), reinforcement through independent interpretation followed by AI-guided debriefing, and a final post-test evaluation. Case difficulty across assessment phases is balanced using a stratified randomization approach to ensure equivalent technical complexity.

Participant performance is evaluated using a predefined 16-item objective scoring system assessing technical validity, numerical parameter interpretation, and diagnostic synthesis. All assessments are independently reviewed by two blinded urologists, with adjudication by a third expert in cases of disagreement. Changes in interpretation accuracy over time are used to quantify the learning curve associated with LLM-assisted education.

All urodynamic data are fully anonymized prior to use, and no patient-identifiable information is shared. Participation is voluntary, and written informed consent is obtained from all residents. The study is conducted following institutional ethical standards and aims to provide evidence for the role of large language models as interactive tutors in advanced medical education.

ELIGIBILITY:
Inclusion Criteria:

Urology residents currently enrolled in an accredited urology training program

No prior formal certification in urodynamic training

Exclusion Criteria:

Prior completion of a formal urodynamic training course

Declining to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Improvement in Urodynamic Interpretation Accuracy | From baseline (pre-test) to post-test (approximately 4 weeks)
  Change in urodynamic interpretation performance measured using a predefined 16-item objective scoring system assessing technical validity, numerical parameter interpretation, and diagnostic synthesis. Scores are compared across pre-test, mid-test, and post-test assessments to evaluate learning curve progression.

CONTACTS AND LOCATIONS:
Overall Officials: Hüseyin Koçakgöl, MD, Principal Investigator — University of Health Sciences, Erzurum City Hospital
Locations (1):
- University of Health Sciences, Erzurum City Hospital, Department of Urology, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study involves a small sample size and focuses on educational performance outcomes. All analyses will be reported in aggregate form without identifiable individual-level data.

REFERENCES:
- [Background] Frigerio M, Barba M, Cola A, Volontè S, Marino G, Regusci L, Sorice P, Ruggeri G, Castronovo F, Serati M, Torella M, Braga A. The Learning Curve of Urodynamics for the Evaluation of Lower Urinary Tract Symptoms. Medicina (Kaunas). 2022 Feb 23;58(3):341. doi: 10.3390/medicina58030341. PMID: 35334517; PMCID: PMC8955767.